CLINICAL TRIAL: NCT03531021
Title: Increasing Heart Healthy Behaviors in Youth With Type 1 Diabetes: A Pilot Study
Brief Title: Increasing Heart Healthy Behaviors in Youth With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joslin Diabetes Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017-34
Record Dates: First submitted 2018-04-26; First posted 2018-05-21 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Type1diabetes; Cardiovascular Risk Factor
Keywords: type 1 diabetes; cardiovascular risk factor; teenager
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Randomized, attention-matched trial with 1:1 randomization at a single center. Subjects will be randomized in two strata, by age (14-16 years and 17-19 years).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heart healthy intervention (Experimental): The intervention group will receive 2 modules (one in in person and one by video conference) and will receive follow-up phone calls/emails by study staff 3 weeks following each visit to review education and strategies for and barriers to reaching goals. Intervention sessions must include teen; parents may attend if they wish. Participants will be placed on teams and encouraged to complete behavioral challenges to earn points towards a cash reward.
  Interventions: Behavioral: Heart healthy intervention
- Attention Control (No Intervention): There will be a delayed intervention for the control group with study handouts after 3 months. The control group will meet with the RAs for demographic and survey completion and receive reminder phone calls/emails in order to match for attention.

INTERVENTIONS:
Behavioral: Heart healthy intervention — Intervention consists of educational modules, goal setting and brainstorming around strategies and barriers, and a series of heart healthy challenges such as walking a certain number of steps or eating healthy foods a certain number of times in a week.
  Arms: Heart healthy intervention

SUMMARY:
This study is evaluating how to encourage teens to engage in heart healthy behaviors such as being more active or eating in a healthy way. Teens will be randomly assigned to either the usual care group or the group with education, goal-setting, and lifestyle challenges with teammates.

DETAILED DESCRIPTION:
Specific Aim: To develop and pilot test a modular intervention to improve heart healthy self-efficacy and behaviors in teens with type 1 diabetes at elevated cardiovascular disease risk.

Intervention Objective: To evaluate the feasibility and efficacy of a psychoeducational and behavioral intervention to improve heart healthy self-efficacy and behaviors in youth with type 1 diabetes (T1D) at elevated cardiovascular disease (CVD) CVD risk.

Secondary Objective: Assess participation in challenges involving healthy eating and physical activity.

Synopsis of Study Design

Study Design: Randomized, attention-matched trial with 1:1 randomization at a single center. Subjects will be randomized in two strata, by age (14-16 years and 17-19 years).

Study Population: Teens with type 1 diabetes.

Intervention: This pilot study involves a 6-month randomized controlled trial (RCT) comparing 2 study conditions, the behavioral intervention vs. an attention control. Youth will be randomized in 2 strata, by age (14-16 years and 17-19 years). Enrollment will end after 60 participants.

The intervention group will receive 2 modules (one in in person and one by video conference) and will receive follow-up phone calls/emails by study staff 3 weeks following each visit to review education and strategies for and barriers to reaching goals. Intervention sessions must include teen; parents may attend if they wish. Challenges will occur every 2 weeks. Participants will be on teams of about 3-5 teens and the teams may change over the course of the intervention due to staggered enrollment. As team members finish the study, newly randomized teammates will be assigned.

There will be a delayed intervention for the control group with study handouts after 3 months. The control group will meet with the research assistants (RAs) for demographic and survey completion and receive reminder phone calls/emails in order to match for attention.

ELIGIBILITY:
Inclusion Criteria:

* Teens ages 14-19 years old with T1D for ≥6 months
* Current patients at Joslin Diabetes Center
* Teens will have dyslipidemia (defined as LDL ≥100 mg/dl, HDL <40 mg/dl or triglycerides ≥130 mg/dl in past year), overweight or obesity (BMI percentile ≥85th at screening), prehypertensive or hypertensive blood pressure on day of screening visit, or A1c ≥8.0%
* Youth and parents must be English speaking, without significant learning disabilities, and intend to continue care at our center.
* Access to a smart phone with video conferencing capabilities

Exclusion Criteria:

* Participation in an interventional study within the past 3 months.
* Unwilling to comply with study procedures
* Prescribed BP and/or lipid-lowering medications (besides over-the-counter supplements)
* Contraindication to exercise

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2018-05-03 (Actual); Primary Completion 2019-02-08 (Actual); Study Completion 2019-02-08 (Actual)

PRIMARY OUTCOMES:
Adolescent Food Habits Checklist | 3 months
  healthy eating questionnaire, 23 question true/false survey, score range from 0-23, higher scores indicate healthier habits, no subscales.

SECONDARY OUTCOMES:
Adiposity | 3 months
  changes in zbmi
Blood pressure | 3 months
  Changes in blood pressure percentile
Changes in lipid levels | 3 months
  Changes in lipid levels from before study until study end
Activity level | 3 months
  Documentation of how active participants were during study
Exercise Confidence Survey | 3 months
  evaluation of self-efficacy for exercise
Healthy Eating Self-Efficacy Survey | 3 months
  healthy eating self-efficacy measure
Eating Habits Confidence Survey | 3 months
  evaluation of how confident participants are that they can eat in a healthy way
Acceptance of medication for CVD risk survey | 3 months
  brief questions to evaluate willingness to take medication if prescribed
Engagement with behavioral challenges | 3 months
  Proportion of intervention participants who completed challenges
Change in weight | 3 months
  change in weight in kg between enrollment and study completion

CONTACTS AND LOCATIONS:
Overall Officials: Lori Laffel, Principal Investigator — Joslin Diabetes Center
Locations (1):
- Joslin Diabetes Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maxwell TK, Charmant CO, Volkening LK, Laffel LM, Katz ML. A Randomized Pilot Trial Using Mobile Health and Financial Incentives to Motivate Heart-Healthy Behaviors in Adolescents With Type 1 Diabetes. J Diabetes Sci Technol. 2023 May;17(3):855-856. doi: 10.1177/19322968231155151. Epub 2023 Feb 23. No abstract available. PMID 36824050